CLINICAL TRIAL: NCT04592952
Title: Hypersensitivity to CGRP as a Predictive Biomarker of Migraine Prevention With Erenumab
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Messoud Ashina, MD, Professor of Neurology, Danish Headache Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-20047793
Record Dates: First submitted 2020-10-06; First posted 2020-10-19 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Calcitonin Gene-Related Peptide; erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm (Experimental): Provocation Phase: Intravenous infusion of 1.5 µg/min of calcitonin-gene related peptide over 20 minutes.
  Open-Label Treatment Phase: Erenumab packed in a SureClick® Autoinjector Pen (AI)
  Interventions: Drug: Calcitonin Gene-Related Peptide; Drug: Erenumab

INTERVENTIONS:
Drug: Calcitonin Gene-Related Peptide — Intravenous infusion of 1.5 µg/min of calcitonin-gene related peptide over 20 minutes.
  Other Names: CGRP
Drug: Erenumab — Erenumab 70 mg or 140 mg packed in a SureClick® Autoinjector Pen (AI)
  Other Names: Aimovig

SUMMARY:
To explore the relationship between clinical response to erenumab and response to intravenous infusion of calcitonin gene-related peptide in individuals with migraine.

DETAILED DESCRIPTION:
This is a single-center, non-randomized, single-arm, open-label study, in which adults with episodic or chronic migraine will receive intravenous infusion with calcitonin gene-related peptide and subsequently be treated with erenumab. The study will consist of the following elements:

* Provocation Phase (1 experimental day with intravenous infusion of calcitonin gene-related peptide)
* Screening/Baseline Phase (4 weeks)
* Open-Label Treatment Phase (24 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age upon entry into screening
* History of migraine with or without aura for ≥ 12 months according to the International Classification of Headache Disorders 3rd Edition (ICHD-3) criteria
* ≥ 4 headache days that meet criteria as migraine days per month on average across the 3 months before screening
* Subject has provided informed consent prior to initiation of any study-specific activities/procedures.
* Must have demonstrated greater than or equal to 75% compliance in Headache Diary usage during the 4-week run-period prior to Day 1 of the open-label treatment phase.

Exclusion Criteria:

* > 50 years of age at migraine onset
* History of cluster headache or hemiplegic migraine
* Inability to differentiate migraine from other headaches
* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behavior
* History or evidence of any other clinically significant disorder, condition or disease that, in the opinion of the site investigator, would pose a risk to subject safety or interfere with study evaluation, procedures or completion
* Previously received erenumab (Aimovig)
* Received anti-CGRP monoclonal antibody within 3 months prior to the CGRP-infusion
* Currently receiving treatment in another investigational device or drug study, or less than 30 days or 5 half-lives since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Female subjects of childbearing potential with a positive pregnancy test during any study visit
* Female subject is pregnant or breastfeeding or planning to become pregnant during the study
* Evidence of current pregnancy or breastfeeding
* Female subject of childbearing potential unwilling to use an acceptable method of effective contraception
* Hypertension on the experimental day defined as systolic blood pressure ≥ 150mmHg or diastolic blood pressure ≥ 100mmHg
* Hypotension on the experimental day defined as systolic blood pressure < 90mmHg or diastolic blood pressure < 50mmHg
* Any headache (including migraine) within 24 hours prior to the start of the CGRP-infusion
* Intake of any analgesics or migraine-specific medications within 24 hours prior to the start of the CGRP-infusion
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or comply with all required study procedures to the best of the subject and study investigator's knowledge

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Headache Diary (Baseline Phase and Treatment Phase) | Baseline Phase (Day -28 to Day 1) to Week 24
  Headache diary with daily entries to record migraine-related data (e.g. migraine days, headache days, number of days with use of acute migraine medication, number of days with aura).

SECONDARY OUTCOMES:
Headache Diary (Provocation Phase) | Provocation Phase (12 Hours)
  Subjects will be instructed to fill out a headache diary during the 12-hour observational period. The diary will be used to record migraine-related data (e.g. location, quality, intensity, aggravation by routine physical activity, use of acute migraine medication, nausea, vomiting, photophobia, and phonophobia)
Semi-Structured Interview | 1 Hour
  In-person semi-structured interview to record migraine-related data (e.g. location, quality, intensity, aggravation by routine physical activity, use of acute migraine medication, nausea, vomiting, photophobia, phonophobia, premonitory symptoms, postdromal symptoms, trigger factors, autonomic symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Copenhagen, Glostrup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Khazali HM, Ashina H, Christensen RH, Wiggers A, Rose K, Iljazi A, Amin FM, Ashina M, Snellman J, Maio-Twofoot T, Schytz HW. Hypersensitivity to CGRP as a predictive biomarker of migraine prevention with erenumab. Cephalalgia. 2024 Jun;44(6):3331024241258734. doi: 10.1177/03331024241258734. PMID 38859744
- [Derived] Al-Khazali HM, Ashina H, Christensen RH, Wiggers A, Rose K, Iljazi A, Schytz HW, Amin FM, Ashina M. An exploratory analysis of clinical and sociodemographic factors in CGRP-induced migraine attacks: A REFORM study. Cephalalgia. 2023 Oct;43(10):3331024231206375. doi: 10.1177/03331024231206375. PMID 37815254
- [Derived] Al-Khazali HM, Ashina H, Wiggers A, Rose K, Iljazi A, Christensen RH, Schytz HW, Amin FM, Ashina M. Calcitonin gene-related peptide causes migraine aura. J Headache Pain. 2023 Sep 7;24(1):124. doi: 10.1186/s10194-023-01656-4. PMID 37679723
- [Derived] Karlsson WK, Ashina H, Cullum CK, Christensen RH, Al-Khazali HM, Amin FM, Ashina M; REFORM Investigators. The Registry for Migraine (REFORM) study: methodology, demographics, and baseline clinical characteristics. J Headache Pain. 2023 Jun 12;24(1):70. doi: 10.1186/s10194-023-01604-2. PMID 37303034